CLINICAL TRIAL: NCT01983449
Title: Delivery of Dexamethasone to the Adventitia to eNhance Clinical Efficacy After Femoropopliteal Revascularization
Brief Title: Effectiveness of Adventitial Dexamethasone in Peripheral Artery Disease
Acronym: DANCE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mercator MedSystems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TSP0149; 1142183 (Other: Western IRB)
Record Dates: First submitted 2013-11-04; First posted 2013-11-14 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Peripheral Arterial Diseases
Keywords: Adventitia; Peripheral Artery Disease; Restenosis; Inflammation; Anti-Inflammatory; Dexamethasone
MeSH Terms: conditions — Peripheral Arterial Disease; Inflammation | interventions — dexamethasone 21-phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adventitial Dexamethasone (Experimental): In patients receiving either angioplasty or atherectomy-based revascularization (pre-stratified to each by 50% of the total study), dexamethasone will be delivered to the adventitia following revascularization.
  Interventions: Drug: Dexamethasone Sodium Phosphate Injection, USP

INTERVENTIONS:
Drug: Dexamethasone Sodium Phosphate Injection, USP — Adventitial infusion of dexamethasone after angioplasty or atherectomy-based revascularization of the superficial femoral or popliteal artery.

SUMMARY:
To assess the safety and effectiveness of adventitial deposition of the Study Drug in reducing inflammation and restenosis in patients with clinical evidence of claudication or critical limb ischemia and an angiographically significant lesion in the superficial femoral and/or popliteal arteries.

Study Drug and Dose: Dexamethasone Sodium Phosphate Injection, USP, 4 mg/ml, with dilute contrast (17%) administered to the adventitia in a dose of 1.6 mg per cm of desired vessel treatment length.

DETAILED DESCRIPTION:
This trial will examine the ability for adventitial dexamethasone to safely delay restenosis in patients at least 18 years of age, who have peripheral atherosclerotic lesions involving the superficial femoral and/or popliteal arteries. These patients have no current therapeutic alternatives beyond the procedure used to open, or revascularize, their superficial femoral and/or popliteal arteries. Metal stents have the potential to fracture when implanted in this artery segment due to continual flexion and bending of the knee. It is desirable to improve the patency of this artery after percutaneous transluminal angioplasty (PTA) and/or atherectomy-based revascularization.

ELIGIBILITY:
Inclusion Criteria:

* Screening Criteria

  * Male or non-pregnant female ≥18 years of age
  * Rutherford Clinical Category 2-4
  * Clinical diagnosis of PAD requiring revascularization, secondary to atherosclerosis affecting a lower limb
  * Patient is willing to provide informed consent and comply with the required follow up visits, testing schedule, and medication regimen
* Procedural Criteria

  * De novo or nonstented restenotic lesions >90 days from prior angioplasty and/or atherectomy, at least 3 cm from any previously placed stent or vascular surgery site
  * >70% diameter stenosis up to 15 cm in total length (with no greater than 3 cm length of contiguous intervening normal artery) in the superficial femoral and/or popliteal artery (between the profunda and tibioperoneal trunk)
  * Reference vessel diameter ≥3mm and ≤ 8mm
  * Successful wire crossing of lesion
  * A patent artery proximal to the index lesion free from significant stenosis (significant stenosis is defined as >50% in iliac or >30% stenosis in common femoral artery) as confirmed by angiography (treatment of target lesion after successful treatment of iliac or common femoral artery lesions is acceptable)

Exclusion Criteria:

* Screening Criteria

  * Pregnant, nursing or planning on becoming pregnant in < 2 years
  * Life expectancy of <2 years
  * Known active malignancy
  * History of solid organ transplantation
  * Patient actively participating in another investigational device or drug study
  * History of hemorrhagic stroke within 3 months
  * Previous or planned surgical or interventional procedure within 30 days of index procedure
  * Chronic renal insufficiency with eGFR <29
  * Prior bypass surgery, stenting of the target lesion
  * Inability to take required study medications
  * Contra-indication or known hypersensitivity to dexamethasone sodium phosphate, contrast media, or Physician prescribed antiplatelet regimen as indicated
  * Systemic fungal infection
  * Anticipated use of IIb/IIIa inhibitor prior to index lesion treatment
  * Acute or sub-acute thrombus, acute vessel occlusion or sudden symptom onset
  * Acute limb ischemia
  * Prior participation of the index limb in the current study (contralateral treatment is allowed)
  * Inability to ambulate (e.g. from prior ipsilateral or contralateral amputation)
  * Patient is receiving steroids already, however locally acting inhaled steroids for asthma treatment do not exclude patients from the trial
* Procedural Criteria

  * Lesions extending into the trifurcation or above the profunda
  * Heavy eccentric or moderate circumferential calcification at index lesion, which in the judgment of the investigator would prevent penetration of the Micro-Infusion Catheter needle through the vessel wall
  * Lesion length is >15 cm as measured from proximal normal vessel to distal normal vessel, or there is no normal proximal arterial segment in which duplex ultrasound velocity ratios can be measured
  * Inadequate distal outflow defined as absence of at least one patent tibial artery (no lesion >50% stenosis) with flow into the foot
  * Use of adjunctive therapies other than angioplasty, atherectomy (mechanical or laser) or bare metal stenting (i.e. scoring/cutting balloon, drug-eluting stent, drug-coated balloon, cryoplasty, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2013-11; Primary Completion 2016-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
MALE-POD | 30 days
  Acute safety safety outcomes will be determined by evaluating the type, frequency, severity, and relatedness of Major Adverse Limb Events or Peri-Operative Death (MALE+POD) within 30 days from the procedure for all subjects.
Duplex ultrasound index lesion binary restenosis | 6 months
  Binary restenosis will be judged by core laboratory interpretation with peak systolic velocity ratio (PSVR) greater than 2.4.
Duplex ultrasound index lesion binary restenosis | 12 months
  Binary restenosis will be judged by core laboratory interpretation with peak systolic velocity ratio (PSVR) greater than 2.4.

SECONDARY OUTCOMES:
Long term safety | 30 days to 6 months
  Long term safety outcomes that occur after 30 days through 6 months post-procedure will be determined by evaluating adverse events.
Duplex ultrasound index lesion flow limiting restenosis | 6 and 12 months
  Flow limiting restenosis will be judged by core laboratory as PSVR>4.0.
Change in inflammatory biomarkers | Baseline and 24 hours
  Change in inflammatory biomarkers will be measured with a panel of biomarkers in 1/3 of patients.
Vascular patency | 6, 12, 18 and 24 months
  Target lesion revascularization (TLR) rate, target extremity revascularization (TER) rate, limb salvage rate and primary patency (PSVR≤2.4 and no TLR) at 6, 12, 18 and 24 months. Note: provisional stenting performed during the index procedure shall not be considered to be TLR, TER or loss of primary patency.
Clinical outcome measures | 1, 6, 12, 18 and 24 months
  Modified Walking Impairment Questionnaire, Ankle-Brachial Index, Rutherford Score.
Infusion Technical Success | Intraprocedural
  Distribution grade around infusion sites.
Procedural Success | Intraprocedural
  Establishment of antegrade flow with residual stenosis of <30% by angiogram.
Healthcare Economics | 30 days
  Number of return visits and hospitalizations, time from index procedure to required revascularization and number of index-lesion-related readmissions within 30 days will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmood Razavi, MD, Principal Investigator — St. Joseph's Vascular Institute
Locations (38):
- United States (38):
  - Arizona Heart Hospital / Abrazo Health Care Research / Tenet Health, Phoenix, Arizona
  - Pima Vascular, Tucson, Arizona
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Cardiovascular Medical Group of Southern California / Cardiovascular Research Foundation, Beverly Hills, California
  - St. Joseph Hospital of Orange Heart and Vascular Center, Orange, California
  - San Francisco VA Medical Center, San Francisco, California
  - University of California San Francisco Medical Center, San Francisco, California
  - VA Eastern Colorado Healthcare System, Denver, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - MedStar Health Washington Hospital Center, Washington D.C., District of Columbia
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Munroe Regional Medical Center, Ocala, Florida
  - Coastal Vascular & Interventional, Pensacola, Florida
  - St. Joseph Hospital, Fort Wayne, Indiana
  - Willis-Knighton Medical Center, Shreveport, Louisiana
  - UMass Medical School, Worcester, Massachusetts
  - St. John Providence Hospital and Medical Center, Detroit, Michigan
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - St.Louis University Hospital, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Deborah Heart & Lung Center, Browns Mills, New Jersey
  - Hunterdon Medical Center, Flemington, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Albany Vascular Group, Albany, New York
  - Gotham Cardiovascular Research / New York Cardiovascular Associates, New York, New York
  - Columbia University Medical Center, New York, New York
  - UNC Health Care - Rex Hospital, Raleigh, North Carolina
  - OhioHealth, Columbus, Ohio
  - UPMC Heart & Vascular Institute, Pittsburgh, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - Wellmont CVA Heart Institute, Kingsport, Tennessee
  - DFW Vascular Group, Dallas, Texas
  - Plaza Medical Center at Fort Worth, Fort Worth, Texas
  - Palestine Regional Medical Center, Palestine, Texas
  - Mission Research Institute (Guadalupe Regional Medical Center), Seguin, Texas
  - Alpine Research / Utah Cardiology, Salt Lake City, Utah
  - University of Washington Veterans Center, Seattle, Washington

REFERENCES:
- [Derived] Razavi MK, Donohoe D, D'Agostino RB Jr, Jaff MR, Adams G; DANCE Investigators. Adventitial Drug Delivery of Dexamethasone to Improve Primary Patency in the Treatment of Superficial Femoral and Popliteal Artery Disease: 12-Month Results From the DANCE Clinical Trial. JACC Cardiovasc Interv. 2018 May 28;11(10):921-931. doi: 10.1016/j.jcin.2017.12.015. Epub 2018 May 2. PMID 29730377